CLINICAL TRIAL: NCT04516096
Title: AMX0035 for Amyotrophic Lateral Sclerosis - Compassionate Use Protocol
Brief Title: A Compassionate Use Protocol of AMX0035 for Treatment of Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A35-003
Record Dates: First submitted 2020-08-09; First posted 2020-08-18 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Intervention Model Description: Open label long term extension of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMX-0035 long term treatment extension (Experimental): AMX0035 administered twice daily p.o.
  Interventions: Drug: AMX0035

INTERVENTIONS:
Drug: AMX0035 — Tauroursodeoxycholic Acid and Sodium Phenylbutyrate orally given twice a day

SUMMARY:
The protocol is intended to provide extended treatment with AMX0035 to patients who previously participated in an Amylyx sponsored study of AMX0035 for ALS.

DETAILED DESCRIPTION:
In this open-label, compassionate extended use study, patients who have completed their participation in an Amylyx sponsored protocol for ALS may be offered compassionate use extension of treatment with AMX0035 under this protocol. Patient currently treated with AMX0035 will continue to receive treatment at their current dose/regimen. Patients who have interrupted AMX0035 for more than 28 days will resume AMX0035 treatment with 1 sachet (oral [or feeding tube]) once a day in the morning to be escalated to twice a day (morning and evening) after approximately 2 weeks on the basis of GI tolerance. Enrolled patients will complete regular outpatient visit approximately every 16 weeks (± 2 weeks). Completion of the ALS functional rating scale (ALSFRS-R) will be optional.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has completed follow-up in an Amylyx sponsored trial of AMX0035 for the treatment of ALS will be eligible to enroll into this Protocol
* Capable of providing informed consent
* Capable and willing to follow trial procedures
* Capable and willing of travelling to the site at regular intervals for interim site visits and to return and collect study drug or able to attend telemedicine remote site visits if such are currently in use at the site
* Participants who have established care with a neurologist at the specialized ALS center involved in the study and will maintain this clinical care throughout the duration of the protocol.
* Women of child bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the study and 3 months after last dose of study drug.
* Women must not be nursing, be pregnant or planning to become pregnant for the duration of the study and 3 months after last dose of study drug
* Men must agree to practice contraception for the duration of the study and 3 months after last dose of study drug. Men must not plan to father a child or provide sperm for donation for the duration of the study and 3 months after last dose of study drug

Exclusion Criteria:

* Ongoing severe adverse events that in the opinion of the Site Investigator are contraindication to the study drug, including severe renal or liver insufficiency or Class III/IV heart failure (per New York Heart Association)
* Ongoing serious adverse event that was assessed as related to study drug per the Site Investigator
* Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the patient to provide informed consent, according to Site Investigator judgment;
* Current severe biliary disease which may result in the investigator medical judgement in biliary obstruction including for example active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gallbladder polyps, gangrene of the gallbladder, abscess of the gallbladder;
* Clinically significant unstable medical condition (other than ALS) that would pose a risk to the patient if they were to participate in the study, according to Site Investigator judgment;
* Treatment, current or within 90 days from screening with any cell therapies or gene therapies;
* Implantation of Diaphragm Pacing System (DPS);
* Current or planned exposure to any prohibited medications listed in Section

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Treatment emergent Adverse Events | Through study completion an average of 1 year
  Rate of treatment emergent adverse events during AMX0035 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Machelle Manual, PhD, Study Director — Amylyx Pharmaceuticals Inc.
Locations (5):
- United States (5):
  - Forbes Norris MDA/ALS Research Center - California Pacific Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina